CLINICAL TRIAL: NCT07082946
Title: Mechanism of Perioperative Systemic Inflammation-Induced Postoperative Neurocognitive Disorders in Chronic Liver Disease Patients Via Blood-Brain Barrier Disruption
Brief Title: Mechanisms of Perioperative Systemic Inflammation in the Development of PND in Cirrhotic Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Peng Li, Principal Investigator, Sichuan Provincial People's Hospital
Other Study IDs: SPPH202360
Record Dates: First submitted 2025-07-06; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples With DNA — blood serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with liver cirrhosis scheduled for upper abdominal surgery
- Patients without liver cirrhosis scheduled for upper abdominal surgery

SUMMARY:
Chronic Liver Disease (CLD) is associated with significant cognitive dysfunction, including hepatic encephalopathy (HE), which is driven by systemic inflammation and blood-brain barrier (BBB) disruption. Perioperative Neurocognitive Disorders (PND), comprising postoperative delirium (POD) and postoperative cognitive dysfunction (POCD), further exacerbate these impairments, particularly in cirrhotic patients undergoing major surgery. However, the mechanisms linking systemic inflammation, BBB dysfunction, and PND remain poorly understood. This study aimed to investigate perioperative cognitive changes and inflammatory markers in cirrhotic and non-cirrhotic patients undergoing major abdominal surgery, and to explore the effects of cirrhosis and surgical intervention on central nervous system inflammation and cognitive dysfunction using a rat model. The investigators conducted a prospective study on cirrhotic and non-cirrhotic patients undergoing major abdominal surgery. Perioperative cognitive function was assessed using validated tools, and inflammatory markers were analyzed using Olink Target protein detection and bioinformatics approaches. Additionally, the investigators established a cirrhosis model using bile duct ligation (CBDL) in rats, followed by exploratory laparotomy to evaluate behavioral performance, BBB integrity and levels of inflammatory cytokines in serum and brain tissue.

DETAILED DESCRIPTION:
Chronic Liver Disease (CLD) is associated with significant cognitive dysfunction, including hepatic encephalopathy (HE), which is driven by systemic inflammation and blood-brain barrier (BBB) disruption. Perioperative Neurocognitive Disorders (PND), comprising postoperative delirium (POD) and postoperative cognitive dysfunction (POCD), further exacerbate these impairments, particularly in cirrhotic patients undergoing major surgery. However, the mechanisms linking systemic inflammation, BBB dysfunction, and PND remain poorly understood. This study aimed to investigate perioperative cognitive changes and inflammatory markers in cirrhotic and non-cirrhotic patients undergoing major abdominal surgery, and to explore the effects of cirrhosis and surgical intervention on central nervous system inflammation and cognitive dysfunction using a rat model. The investigators conducted a prospective study on cirrhotic and non-cirrhotic patients undergoing major abdominal surgery. Perioperative cognitive function was assessed using validated tools, and inflammatory markers were analyzed using Olink Target protein detection and bioinformatics approaches. Additionally, the investigators established a cirrhosis model using bile duct ligation (CBDL) in rats, followed by exploratory laparotomy to evaluate behavioral performance, BBB integrity and levels of inflammatory cytokines in serum and brain tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-80 years
2. Patients with or without liver cirrhosis scheduled for upper abdominal surgery due to various clinical indications
3. Ability to comply with the study protocol and provide informed consent

Exclusion Criteria:

1. Comorbid severe cardiac, pulmonary, or renal diseases
2. Patients with mental status incompatible with study participation, including:

   * Psychiatric disorders
   * Inability to communicate clearly
3. Any condition preventing effective communication or cooperation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients scheduled for surgical treatment at Sichuan Provincial People's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative delirium within 7 days after upper abdominal surgery in patients with liver cirrhosis | within 7 days after sugery

SECONDARY OUTCOMES:
The incidence of postoperative delirium within 7 days after upper abdominal surgery in patients without liver cirrhosis | within 7 days after sugery

IPD SHARING:
Plan to Share IPD: Undecided